CLINICAL TRIAL: NCT02172950
Title: A Phase III Open Label, Multicenter, Extension Study to Assess the Safety and Efficacy of Recombinant Coagulation Factor VIII (rVIII-SingleChain, CSL627) in Subjects With Severe Hemophilia A
Brief Title: An Open-label Safety and Efficacy Study of Recombinant FVIII in Patients With Severe Hemophilia A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSL627_3001; 2013-003262-13 (EudraCT Number)
Record Dates: First submitted 2014-06-23; First posted 2014-06-24 (Estimated); Results first posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-09

CONDITIONS: Hemophilia A; Severe Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Previously treated patients (PTPs) (Experimental): The investigator will assign subjects to either prophylaxis or on-demand treatment regimens for rVIII-SingleChain by intravenous injection. The investigator will determine the rVIII-SingleChain dose and dosing schedule for the subject based upon the subject's pharmacokinetic (PK) profile, rVIII-SingleChain PK data, previous FVIII treatment regimen, and bleeding phenotype, if available.
  Interventions: Biological: rVIII-SingleChain
- Previously untreated patients (PUPs) (Experimental): The investigator will assign subjects to either prophylaxis or on-demand treatment regimens for rVIII-SingleChain by intravenous injection. The investigator will determine the rVIII-SingleChain dose and dosing schedule at their discretion, taking into consideration the World Federation of Hemophilia (WFH) guidelines, the type of bleeding episode, location of the bleeding, subject's age, and other disease characteristics.
  Interventions: Biological: rVIII-SingleChain

INTERVENTIONS:
Biological: rVIII-SingleChain — Recombinant single-chain coagulation factor VIII
  Other Names: CSL627

SUMMARY:
This multicenter, open-label, phase 3 extension study will investigate the safety and efficacy of rVIII-SingleChain for prophylaxis and on-demand treatment of bleeding episodes in at least 200 previously treated patients (PTPs) with severe congenital hemophilia A and previous exposure to FVIII products who achieve at least 100 exposure days (EDs) to rVIII-SingleChain in this study, as well as in previously untreated patients (PUPs) with no previous exposure to any FVIII product who achieve at least 50 EDs to rVIII-SingleChain in this study. A substudy (open to both PTPs and PUPs) will investigate the use of rVIII-SingleChain in surgery. A substudy (open to PUPs who develop an inhibitor to rVIII-SingleChain) will investigate the use of rVIII-SingleChain in immune tolerance induction (ITI) therapy.

ELIGIBILITY:
Inclusion Criteria:

PTPs:

* Males of any age who have been diagnosed with severe congenital hemophilia A (FVIII activity levels < 1%) and who participated in a previous CSL-sponsored clinical study with rVIII-SingleChain.
* Males 0 to <65 years age who have been diagnosed with severe congenital hemophilia A (FVIII activity levels < 1%), who have at least 50 EDs to any FVIII product, and who are not currently enrolled in a CSL-sponsored clinical study with rVIII-SingleChain.

PUPs:

* Males 0 to <18 years of who have been diagnosed with severe congenital hemophilia A (FVIII activity levels < 1%)
* No prior exposure to any Factor VIII product (with the exception of short-term use of blood products).

ITI substudy:

* PUPs who have developed a confirmed inhibitor to rVIII-SingleChain in the main study.

Exclusion Criteria:

* Known or suspected hypersensitivity to rVIII-SingleChain or to any excipients of rVIII-SingleChain or Chinese hamster ovary (CHO) proteins.
* Currently receiving a therapy not permitted during the study.
* Serum creatinine > 2 x upper limit of normal, alanine aminotransferase or aspartate aminotransferase > 5 x upper limit of normal at Screening (if specified)
* Any first-order family (eg, siblings) history of FVIII inhibitors
* For PTPs not rolling over directly from a CSL-sponsored clinical study with rVIII-SingleChain: any history of or current FVIII inhibitors

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2014-10-13; Primary Completion 2021-01-19 (Actual); Study Completion 2021-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Program Director, Study Director — CSL Behring
Locations (64):
- United States (9):
  - Study Site 8400213, San Diego, California
  - Study Site 8400241, Aurora, Colorado
  - Study Site 8400118, Hartford, Connecticut
  - Study Site 8400116, Miami, Florida
  - Study Site 8400184, Chicago, Illinois
  - Study Site 8400204, New Orleans, Louisiana
  - Study Site 8400240, Dallas, Texas
  - Study Site 8400041, Houston, Texas
  - Study Site 8400154, Milwaukee, Wisconsin
- Australia (3):
  - Study Site 0360014, Melbourne
  - Study Site 0360028, Nedlands
  - Study Site 0360031, Perth
- Austria (4):
  - Study Site 0400012, Graz
  - Study Site 0400003, Linz
  - Study Site 0400001, Vienna
  - Study Site 0400002, Vienna
- Study Site 1240022, Saint John, Canada
- Study Site 2030017, Hradec Králové, Czechia
- France (5):
  - Study Site 2500015, Brest
  - Study Site 2500017, Le Kremlin-Bicêtre
  - Study Site 2500028, Lille
  - Study Site 2500018, Nantes
  - Study Site 2500002, Paris
- Study Site 2680001, Tbilisi, Georgia
- Germany (4):
  - Study Site 2760034, Bonn
  - Study Site 2760091, Frankfurt
  - Study Site 2760087, Giessen
  - Study Site 2760066, Hanover
- Study Site 3480007, Debrecen, Hungary
- Study Site 3720002, Dublin, Ireland
- Study Site 3800023, Milan, Italy
- Japan (5):
  - Study Site 3920031, Hyōgo
  - Study Site 3920029, Nagoya
  - Study Site 3920064, Okayama
  - Study Site 3920033, Saitama
  - Study Site 3920025, Tokyo
- Study Site 4220007, Beirut, Lebanon
- Study Site 4580001, Kuala Lumpur, Malaysia
- Netherlands (3):
  - Study Site 5280006, Amsterdam-Zuidoost
  - Study Site 5280008, Nijmegen
  - Study Site 5280007, Utrecht
- Philippines (2):
  - Study Site 6080001, Cebu City
  - Study Site 6080002, Davao City
- Poland (4):
  - Study Site 6160013, Gdansk
  - Study Site 6160038, Krakow
  - Study Site 6160035, Rzeszów
  - Study Site 6160014, Wroclaw
- Study Site 6200001, Porto, Portugal
- Romania (2):
  - Study Site 6420030, Bucharest
  - Study Site 6420037, Timișoara
- Study Site 7100001, Parktown, South Africa
- Spain (4):
  - Study Site 7240008, A Coruña
  - Study Site 7240021, Barcelona
  - Study Site 7240007, Madrid
  - Study Site 7240023, Valencia
- Study Site 7560010, Lucerne, Switzerland
- Thailand (5):
  - Study Site 7640001, Bangkok
  - Study Site 7640005, Bangkok
  - Study Site 7640002, Chiang Mai
  - Study Site 7640004, Khon Kaen
  - Study Site 7640003, Songkhla
- Ukraine (2):
  - Study Site 8040007, Dnipropetrovsk
  - Study Site 8040005, Lviv
- Study Site 8260008, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Previously Treated Patients (PTPs) | Previously Untreated Patients (PUPs)
Started | 222 | 24
Completed | 197 | 19
Not Completed | 25 | 5
Not completed — Physician Decision | 3 | 3
Not completed — Lack of Efficacy | 1 | 0
Not completed — Adverse Event | 4 | 1
Not completed — Withdrawal by Subject | 10 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 1 | 0
Not completed — Patient traveling | 1 | 0
Not completed — Patient went to other country | 1 | 0
Not completed — Patient relocated overseas | 1 | 1
Not completed — Patient moving | 1 | 0

BASELINE CHARACTERISTICS:
Population: Age was analyzed separately as PTPs and PUPs
Groups:
- Total: Total of all reporting groups
Arm/Group | Previously Treated Patients (PTPs) | Previously Untreated Patients (PUPs) | Total
Number analyzed (Participants) | 222 | 24 | 246
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 95 | 24 | 119
  Between 18 and 65 years | 126 | 0 | 126
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age was analyzed separately as PTPs and PUPs
  years
    PTPs: number analyzed (Participants) | 222 | 0 | 222
    PTPs | 22.5 (14.55) |  | 22.5 (14.55)
    PUPs: number analyzed (Participants) | 0 | 24 | 24
    PUPs |  | 1.4 (1.18) | 1.4 (1.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 222 | 24 | 246
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 1 | 11
  Not Hispanic or Latino | 212 | 23 | 235
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 50 | 2 | 52
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 7 | 19
  White | 158 | 15 | 173
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  Czechia | 2 | 0 | 2
  United States | 21 | 1 | 22
  Malaysia | 13 | 2 | 15
  Thailand | 10 | 0 | 10
  Portugal | 2 | 3 | 5
  Austria | 6 | 0 | 6
  Netherlands | 9 | 3 | 12
  Ireland | 5 | 0 | 5
  Poland | 36 | 0 | 36
  France | 7 | 0 | 7
  Romania | 4 | 0 | 4
  Hungary | 2 | 0 | 2
  Japan | 7 | 0 | 7
  Philippines | 18 | 0 | 18
  Ukraine | 17 | 0 | 17
  United Kingdom | 1 | 0 | 1
  Switzerland | 1 | 0 | 1
  Spain | 6 | 0 | 6
  Lebanon | 9 | 3 | 12
  Canada | 1 | 0 | 1
  Italy | 5 | 4 | 9
  South Africa | 14 | 8 | 22
  Georgia | 5 | 0 | 5
  Australia | 11 | 0 | 11
  Germany | 10 | 0 | 10

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Inhibitor Formation to FVIII in Previously Treated Patients (PTPs) With 100 Exposure Days (EDs) to CSL627
Time Frame: At the closest visit after 100 EDs (up to 5 years).
Population: Safety population (SP) - comprised all the Enrolled Population who received at least 1 dose of rVIII-SingleChain (CSL627) during the study for any reason.
Measure: Number; unit: percentage of paticipants
Groups:
- CSL627: Previously Treated Patients (PTPs): The investigator will assign subjects to either prophylaxis or on-demand treatment regimens for rVIII-SingleChain by intravenous injection. The investigator will determine the rVIII-SingleChain dose and dosing schedule for the subject based upon the subject's pharmacokinetic (PK) profile, rVIII-SingleChain PK data, previous FVIII treatment regimen, and bleeding phenotype, if available.
  rVIII-SingleChain: Recombinant single-chain coagulation factor VIII
Arm/Group | CSL627: Previously Treated Patients (PTPs)
Number analyzed (Participants) | 198
percentage of paticipants | 0

2. Primary Outcome: Number of Previously Untreated Patients (PUPs) With High-titer Inhibitor Formation to FVIII With at Least 50 EDs to CSL627
Description: High-titer inhibitor is defined as an inhibitor titer of ≥ 5 Bethesda units/mL.
Time Frame: At the closest visit after 50 EDs (up to 5 years).
Population: SP
Measure: Number; unit: participants
Groups:
- CSL627: Previously Untreated Patients (PUPs): The investigator will assign subjects to either prophylaxis or on-demand treatment regimens for rVIII-SingleChain by intravenous injection. The investigator will determine the rVIII-SingleChain dose and dosing schedule at their discretion, taking into consideration the World Federation of Hemophilia (WFH) guidelines, the type of bleeding episode, location of the bleeding, subject's age, and other disease characteristics.
  rVIII-SingleChain: Recombinant single-chain coagulation factor VIII
Arm/Group | CSL627: Previously Untreated Patients (PUPs)
Number analyzed (Participants) | 24
participants | 5

3. Primary Outcome: Percent Treatment Success for Major Bleeding Episodes in PUPs
Description: Percentage of major bleeding episodes treated successfully where treatment success for a bleeding episode is defined as a rating of "excellent" or "good" on the investigator's clinical assessment of hemostatic efficacy 4-point scale "excellent, good, moderate or poor/no response". Major bleeding episodes are defined as bleeding episodes for which a subject is required to seek treatment at the hemophilia center or that threatens the subject's life or loss of limb.
Time Frame: Up to 5 years
Population: Efficacy population (EP) - comprised all subjects in the Safety Population who received at least 1 dose of rVIII-SingleChain (CSL627) for either routine prophylaxis treatment or on-demand treatment during the study. This endpoint was analyzed for PUPs only.
Measure: Number; unit: percentage of treatment success
Units Other Than Participants: Major bleeds
Arm/Group | CSL627: Previously Untreated Patients (PUPs)
Number analyzed (Participants) | 23
Number analyzed (Major bleeds) | 1
percentage of treatment success | 100

4. Primary Outcome: Annualized Spontaneous Bleeding Rate in PUPs
Description: The annualized spontaneous bleeding rate for PUPs taking prophylaxis and on-demand treatment regimens.
Time Frame: Up to 5 years
Population: EP. This endpoint was analyzed for PUPs only.
Measure: Mean (Standard Deviation); unit: Number of Spontaneous bleeds per year
Arm/Group | CSL627: Previously Untreated Patients (PUPs)
Number analyzed (Participants) | 23
Number of Spontaneous bleeds per year
  On-demand: number analyzed (Participants) | 12
  On-demand | 1.9 (2.252)
  Prophylaxis | 4.04 (6.374)

5. Secondary Outcome: Percentage of Bleeding Episodes Treated Successfully in PTPs
Description: Percentage of bleeding episodes treated successfully where treatment success for a bleeding episode is defined as a rating of "excellent" or "good" on the investigator's clinical assessment of hemostatic efficacy 4-point scale "excellent, good, moderate or poor/no response".
Time Frame: Up to 5 years
Population: EP
Measure: Number (99% Confidence Interval); unit: Percentage of treated bleeding events
Units Other Than Participants: Number of treated bleeding events
Arm/Group | CSL627: Previously Treated Patients (PTPs)
Number analyzed (Participants) | 222
Number analyzed (Number of treated bleeding events) | 2413
Percentage of treated bleeding events | 87.1 [75.3 to 93.7]

6. Secondary Outcome: Annualized Bleeding Rate in PTPs and PUPs
Description: The annualized bleeding rate for PTPs and PUPs taking prophylaxis and on-demand treatment regimens
Time Frame: Up to 5 years
Population: EP
Measure: Mean (Standard Deviation); unit: Number of bleeds per year
Arm/Group | CSL627: Previously Treated Patients (PTPs) | CSL627: Previously Untreated Patients (PUPs)
Number analyzed (Participants) | 222 | 23
Number of bleeds per year
  On-demand: number analyzed (Participants) | 11 | 10
  On-demand | 28.32 (29.014) | 5.12 (5.331)
  Prophylaxis: number analyzed (Participants) | 209 | 23
  Prophylaxis | 2.84 (4.981) | 5.94 (7.705)

7. Secondary Outcome: Percentage of Bleeding Episodes Requiring 1, 2, 3, or > 3 Injections of CSL627 to Achieve Hemostasis in PTPs and PUPs
Time Frame: Up to 5 years
Population: EP
Measure: Number; unit: Percentage of treated bleeds
Units Other Than Participants: Treated bleeds
Arm/Group | CSL627: Previously Treated Patients (PTPs) | CSL627: Previously Untreated Patients (PUPs)
Number analyzed (Participants) | 222 | 24
Number analyzed (Treated bleeds) | 2413 | 315
Percentage of treated bleeds
  1 infusion | 71.5 | 77.5
  2 infusions | 14.8 | 11.4
  3 infusions | 6.9 | 5.4
  >3 infusions | 6.3 | 3.5

8. Secondary Outcome: Mean Number of On-demand Infusions of CSL627
Time Frame: Up to 5 years
Population: EP. This endpoint analyzes PTPs and PUPs that received on-demand treatment.
Measure: Mean (Standard Deviation); unit: Number of infusions
Arm/Group | CSL627: Previously Treated Patients (PTPs) | CSL627: Previously Untreated Patients (PUPs)
Number analyzed (Participants) | 11 | 12
Number of infusions
  per participant per month | 6.26 (4.778) | 1.23 (1.296)
  per participant per year | 75.18 (57.335) | 14.75 (15.547)

9. Secondary Outcome: Mean On-demand Dose Administered of CSL627
Time Frame: Up to 5 years
Population: EP. This endpoint analyzes PTPs and PUPs that received on-demand treatment.
Measure: Mean (Standard Deviation); unit: IU/kg
Arm/Group | CSL627: Previously Treated Patients (PTPs) | CSL627: Previously Untreated Patients (PUPs)
Number analyzed (Participants) | 11 | 12
IU/kg
  per participant per month | 210.39 (188.106) | 41.93 (44.643)
  per participant per year | 2524.69 (2257.278) | 503.16 (535.712)

10. Secondary Outcome: Mean Prophylaxis Dose Administered of CSL627
Time Frame: Up to 5 years
Population: EP. This endpoint analyzes PTPs and PUPs that received prophylaxis treatment.
Measure: Mean (Standard Deviation); unit: IU/kg
Arm/Group | CSL627: Previously Treated Patients (PTPs) | CSL627: Previously Untreated Patients (PUPs)
Number analyzed (Participants) | 211 | 23
IU/kg
  per participant per month | 380.95 (130.079) | 389.30 (243.191)
  per participant per year | 4571.35 (1560.944) | 4671.54 (2918.288)

11. Secondary Outcome: Mean Total Amount of CSL627 Administered During Surgery Period in PTPs
Time Frame: Day of surgery up to 336 hours post-surgery
Population: Surgery population
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | CSL627: Previously Treated Patients (PTPs)
Number analyzed (Participants) | 24
IU | 51663.0 (62033.25)

12. Secondary Outcome: Total Amount of CSL627 Administered During Surgery Period in PUPs
Time Frame: Day of surgery up to 336 hours post-surgery
Population: Surgery population
Measure: Number; unit: IU
Arm/Group | CSL627: Previously Untreated Patients (PUPs)
Number analyzed (Participants) | 3
IU
  Participant 1 | 15693
  Participant 2 | 5631
  Participant 3 | 7330

13. Secondary Outcome: Hemostatic Efficacy of rVIII-SingleChain for PTPs and PUPs Who Undergo Surgery
Description: The investigator will rate the efficacy of the rVIII-SingleChain treatment during surgery based on a hemostatic efficacy four point rating scale of "excellent, good, moderate or poor/no response".
Time Frame: From the start of surgery through the post-operative recovery (generally up to 14 days after surgery)
Population: Surgery population - comprised all subjects in the Safety Population who received at least 1 dose of rVIII-SingleChain for surgical prophylaxis
Measure: Number; unit: Number of surgeries
Units Other Than Participants: Surgeries
Arm/Group | CSL627: Previously Treated Patients (PTPs) | CSL627: Previously Untreated Patients (PUPs)
Number analyzed (Participants) | 24 | 3
Number analyzed (Surgeries) | 32 | 3
Number of surgeries
  Excellent | 28 | 3
  Good | 4 | 0
  Moderate | 0 | 0
  Poor/No response | 0 | 0

14. Secondary Outcome: Incidence of Inhibitor Formation to FVIII in PTPs After 10 EDs and After 50 EDs
Time Frame: Up to 5 years
Population: SP
Measure: Number; unit: percentage of participants
Arm/Group | CSL627: Previously Treated Patients (PTPs)
Number analyzed (Participants) | 198
percentage of participants
  after 10 EDs | 0
  after 50 EDs | 0

15. Secondary Outcome: Percentage of PTPs and PUPs Developing Antibodies Against CSL627
Time Frame: PTPs: At the closest visit after 100 EDs (up to 5 years). PUPs: At the closest visit after 50 EDs (up to 5 years).
Population: SP
Measure: Number; unit: percentage of participants
Arm/Group | CSL627: Previously Treated Patients (PTPs) | CSL627: Previously Untreated Patients (PUPs)
Number analyzed (Participants) | 222 | 24
percentage of participants | 15.3 | 70.8

16. Secondary Outcome: Percentage of PTPs and PUPs Developing Antibodies to Chinese Hamster Ovary (CHO) Proteins
Time Frame: PTPs: At the closest visit after 100 EDs (up to 5 years). PUPs: At the closest visit after 50 EDs (up to 5 years).
Population: SP
Measure: Number; unit: percentage of participants
Arm/Group | CSL627: Previously Treated Patients (PTPs) | CSL627: Previously Untreated Patients (PUPs)
Number analyzed (Participants) | 222 | 24
percentage of participants | 0 | 0

17. Secondary Outcome: Number of PUPs With High-titer Inhibitor Formation to FVIII After 10 EDs With CSL627
Description: High-titer inhibitor is defined as an inhibitor titer of ≥ 5 Bethesda units/mL.
Time Frame: At the closest visit after 10 EDs (up to 5 years)
Population: SP
Measure: Number; unit: participants
Arm/Group | CSL627: Previously Untreated Patients (PUPs)
Number analyzed (Participants) | 24
participants | 4

18. Secondary Outcome: Number of PUPs With Low-titer Inhibitor Formation to FVIII After 10 EDs and After 50 EDs With CSL627
Description: Low-titer inhibitor is defined as an inhibitor titer of less than 5 Bethesda units/mL.
Time Frame: At the closest visit after 10 and after 50 EDs (up to 5 years)
Population: SP
Measure: Number; unit: participants
Arm/Group | CSL627: Previously Untreated Patients (PUPs)
Number analyzed (Participants) | 24
participants
  after 10 EDs | 4
  after 50 EDs | 0

19. Secondary Outcome: Incidence of Total Inhibitor Formation to FVIII in PUPs
Time Frame: Up to 5 years
Population: SP
Measure: Number; unit: percentage of participants
Arm/Group | CSL627: Previously Untreated Patients (PUPs)
Number analyzed (Participants) | 24
percentage of participants | 50.0

20. Secondary Outcome: Percent Treatment Success for Non-major Bleeding Episodes in PUPs
Description: Percentage of bleeding episodes treated successfully where treatment success for a bleeding episode is defined as a rating of "excellent" or "good" on the investigator's clinical assessment of hemostatic efficacy 4-point scale "excellent, good, moderate or poor/no response". Non-major bleeding episodes are those not requiring treatment at the hemophilia center or not threatening subject's life or loss of limb.
Time Frame: Up to 5 years
Population: EP. This endpoint was analyzed for PUPs only.
Measure: Number (95% Confidence Interval); unit: percentage of treated bleeding events
Units Other Than Participants: Treated bleeding events
Arm/Group | CSL627: Previously Untreated Patients (PUPs)
Number analyzed (Participants) | 24
Number analyzed (Treated bleeding events) | 315
percentage of treated bleeding events | 92.1 [87.0 to 95.3]

21. Secondary Outcome: Percentage of PUPs With Clinically Significant Abnormal Vital Signs Values After First Infusion of CSL627
Description: Vital signs assessments include heart rate, blood pressure, and body temperature. Clinical significance of an abnormality will be assessed by the investigator.
Time Frame: Up to 6 hours after first infusion
Population: SP. This endpoint was analyzed for PUPs only.
Measure: Number; unit: percentage of participants
Arm/Group | CSL627: Previously Untreated Patients (PUPs)
Number analyzed (Participants) | 24
percentage of participants | 0

22. Secondary Outcome: Percentage of PUPs With Treatment-emergent Clinically Significant Abnormal Vital Signs Values
Description: as for outcome 21
Time Frame: Up to 5 years
Population: SP. This endpoint was analyzed for PUPs only.
Measure: Number; unit: percentage of participants
Arm/Group | CSL627: Previously Untreated Patients (PUPs)
Number analyzed (Participants) | 24
percentage of participants | 0

ADVERSE EVENTS:
Time Frame: Up to 5 years
Arm/Group | CSL627: Previously Treated Patients (PTPs) | CSL627: Previously Untreated Patients (PUPs)
All-Cause Mortality (participants affected / at risk) | 1/222 | 0/24
Serious Adverse Events (participants affected / at risk) | 23/222 | 14/24
Other Adverse Events (participants affected / at risk) | 130/222 | 23/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CSL627: Previously Treated Patients (PTPs) (N=222) | CSL627: Previously Untreated Patients (PUPs) (N=24)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Vasospasm (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Abdominal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anti factor VIII antibody positive (Investigations) | 0 (0) | 6 (6)
Inhibiting antibodies positive (Investigations) | 0 (0) | 5 (5)
Factor VIII inhibition (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pregnancy of partner (Social circumstances) | 1 (1) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Lennox-Gastaut syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Blindness transient (Eye disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Haemophilic arthropathy (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendinous contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Acinetobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CSL627: Previously Treated Patients (PTPs) (N=222) | CSL627: Previously Untreated Patients (PUPs) (N=24)
Haematoma (Vascular disorders) | 2 (2) | 2 (3)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 2 (5)
Pyrexia (General disorders) | 14 (18) | 15 (44)
Malaise (General disorders) | 0 (0) | 2 (4)
Fall (Injury, poisoning and procedural complications) | 11 (12) | 3 (5)
Head injury (Injury, poisoning and procedural complications) | 11 (11) | 1 (3)
Contusion (Injury, poisoning and procedural complications) | 11 (13) | 0 (0)
Coronavirus test positive (Investigations) | 0 (0) | 2 (2)
Inhibiting antibodies positive (Investigations) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (19) | 6 (13)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (3)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (3) | 3 (3)
Headache (Nervous system disorders) | 20 (29) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 4 (4) | 2 (2)
Dental caries (Gastrointestinal disorders) | 11 (11) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 5 (6)
Vomiting (Gastrointestinal disorders) | 4 (5) | 3 (8)
Rash (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (3)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 (28) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (2)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2)
Nasopharyngitis (Infections and infestations) | 40 (73) | 9 (15)
Upper respiratory tract infection (Infections and infestations) | 25 (37) | 7 (18)
Influenza (Infections and infestations) | 14 (16) | 4 (6)
Tonsillitis (Infections and infestations) | 13 (17) | 5 (5)
Rhinitis (Infections and infestations) | 7 (7) | 6 (10)
Ear infection (Infections and infestations) | 5 (8) | 5 (9)
Conjunctivitis (Infections and infestations) | 6 (6) | 3 (4)
Bronchitis (Infections and infestations) | 5 (7) | 3 (3)
Varicella (Infections and infestations) | 2 (2) | 6 (7)
Otitis media (Infections and infestations) | 3 (5) | 4 (5)
Viral rhinitis (Infections and infestations) | 1 (1) | 2 (2)
Scarlet fever (Infections and infestations) | 0 (0) | 2 (2)
Tinea capitis (Infections and infestations) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CSL agreements and restrictions on publishing may vary with individual investigators; however, CSL will not prohibit any investigator from publishing. CSL supports the publication of results from all centers of a multi-center trial and generally requires that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-05-26): https://cdn.clinicaltrials.gov/large-docs/50/NCT02172950/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-02): https://cdn.clinicaltrials.gov/large-docs/50/NCT02172950/SAP_001.pdf